CLINICAL TRIAL: NCT01660451
Title: Open-label, Uncontrolled Phase II Trial of Intravenous PI3K Inhibitor BAY80-6946 in Patients With Relapsed, Indolent or Aggressive Non-Hodgkin's Lymphomas
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16349; 2012-002602-52 (EudraCT Number)
Record Dates: First submitted 2012-08-06; First posted 2012-08-08 (Estimated); Results first posted 2018-01-08 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-06

CONDITIONS: Lymphoma, Non-Hodgkin
Keywords: Clinical trial, phase II; Phosphatidylinositol 3-Kinase; Class I, Non-Hodgkin's lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — copanlisib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Copanlisib (indolent NHL) (Experimental): Part A: Participants in this arm will be patients with indolent NHL.
  Interventions: Drug: Copanlisib (Aliqopa, BAY80-6946)
- Copanlisib (aggressive NHL) (Experimental): Part A: Participants in this arm will be patients with aggressive NHL.
  Interventions: Drug: Copanlisib (Aliqopa, BAY80-6946)
- Copanlisib (indolent B-cell NHL) (Experimental): Part B: Participants in this arm will be patients with indolent B-cell NHL.
  Interventions: Drug: Copanlisib (Aliqopa, BAY80-6946)

INTERVENTIONS:
Drug: Copanlisib (Aliqopa, BAY80-6946) — BAY 80-6946 is administered in a normal saline solution, 100 mL, intravenously over 1h. No intravenous glucose preparations should be administered on the days of infusion. Dosing is weekly for the first 3 weeks (on Days 1, 8, and 15) of a 28-day cycle, followed by a 1-week break (i.e., no infusion on Day 22).
  Part A: The individual dose will be 0.8 mg/kg (max. 65 mg) per infusion from Cycle 1 on. The maximum dose of 65 mg should never be exceeded.
  Part B: The individual dose will be 60 mg per infusion from Cycle 1 on.

SUMMARY:
The objective of the study (part A) is to evaluate the efficacy and safety of BAY80-6946 in patients with indolent or aggressive Non-Hodgkin's Lymphoma, who have progressed after standard therapy. 30 patients will be enrolled to both indolent and aggressive disease group. The objective of the study part B (CHRONOS-1) is to evaluate the efficacy and safety of BAY80-6946 in patients with relapsed/refractory follicular lymphoma. 120 patients will be enrolled in the part B of the study. Further objectives are to evaluate the pharmacokinetics and biomarkers. Quality of life will be a further objective of part B of the study.

In a cohort of 20 patients (enrolled both in part A and B) an ECG substudy will be performed to assess the potential for cardiac toxicity and QT/QTc interval prolongation of BAY80-6946.

After an up to 28-day screening period, eligible patients will start treatment with BAY80-6946 at a dose of 0.8 mg/kg (Part A) and at a dose of 60 mg (Part B).

Treatment will be continued until disease has progressed or until another criterion is met for withdrawal from study. An end-of-treatment visit will be performed within 7 days after discontinuation of study treatment. Thirty to 35 days after last study drug administration, a safety followup visit will be performed for the collection of adverse events (AEs) and concomitant medication data. Patients will be contacted quarterly to determine overall survival status up to 4 years after last patient completed treatment. Patients who discontinue study drug for reasons other than disease progression will enter the Active Assessment Follow-up period. The end of study notification to Health Authorities will be based on the completion of the collection of survival data.

The efficacy is measured by the decrease in tumor size. Tumor assessments will be done at Screening, every 8 weeks during Year 1, every 12 weeks during Year 2, and every 6 months during Year 3. Blood samples will be collected for pharmacokinetic analysis. Archival tumor tissue and blood samples will be collected for biomarker analysis (mandatory) and for central pathology review (part B), fresh biopsy tissue will also be collected if available.

ELIGIBILITY:
Inclusion Criteria:

* Indolent NHL:

  * Histologically confirmed diagnosis of follicular lymphoma (FL) grades 1, 2 or 3a, marginal zone lymphoma (including nodal or splenic marginal zone B-cell lymphoma and mucosa-associated lymphoid tissue [MALT] lymphoma), lymphoplasmacytic lymphoma/Waldenström macroglobulinemia, chronic lymphocytic leukemia (CLL).
  * Relapsed after ≥ 2 prior chemotherapy- or immunotherapy-based regimens for indolent NHL, or refractory to 2 prior chemotherapy and/ or immunotherapy-based regimens.
* Aggressive NHL:

  * Histologically confirmed diagnosis of grade 3b follicular lymphoma (FL), transformed indolent lymphoma, diffuse large B-cell lymphoma (DLBCL), mediastinal large B-cell lymphoma, mantle cell lymphoma (MCL), peripheral T-cell lymphoma unspecified, or anaplastic large cell lymphoma primary systemic type, or angioimmunoblastic T cell lymphoma.
  * Relapsed after ≥ 2 prior chemotherapy regimens, including the following: First-line treatment with standard anthracycline-containing regimen (e.g., cyclophosphamide, doxorubicin, vincristine, and prednisone or equivalent). At least 1 additional combination chemotherapy regimen. Patients relapsed after or refractory to first prior chemotherapy- and/or immunotherapy-based regimen for aggressive NHL and not eligible for high-dose regimen followed by transplant. High-dose chemotherapy, or chemoradiotherapy with autologous stem cell transplantation is considered 1 regimen. Patients with CD20 expressing neoplastic cells must have received prior rituximab, if available.
  * Patients with transformed indolent lymphoma must have received at least 2 prior chemotherapy- and/or immunotherapy-based regimens
  * Consent to provide fresh tumor tissue during screening
* Indolent B-cell NHL lymphoma (study part B):

  * Histologically confirmed diagnosis of indolent B-cell NHL, with histological subtype limited to the following:

    * Follicular lymphoma (FL) grade 1-2-3a
    * Small lymphocytic lymphoma (SLL) with absolute lymphocyte count < 5 x 109/L at the time of diagnosis and at study entry
    * Lymphoplasmacytoid lymphoma/Waldenström macroglobulinemia (LPL/WM)
    * Marginal zone lymphoma (MZL) (splenic, nodal, or extranodal)
  * Relapsed or refractory after ≥ 2 prior lines of therapy (refractory defined as not responding to a standard regimen or progressing within 6 months of the last course of a standard regimen). Patients must have received Rituximab and alkylating agents.
* For all patients:

  * Male or female patients > 18 years of age
  * ECOG performance status ≤ 2 (ECOG: Eastern Cooperative Oncology Group)
  * Life expectancy of at least 3 months
  * Adequate bone marrow, liver and renal function as assessed within 7 days before starting study treatment
  * Left ventricular ejection fraction (LVEF) ≥ lower limit of normal (LLN) for the Institution
  * Availability of archival tumor tissue

Exclusion Criteria:

* Uncontrolled hypertension (blood pressure ≥ 150/90 mmHg despite optimal medical management)
* Patients with evidence or history of bleeding diathesis. Any hemorrhage or bleeding event ≥ CTCAE Grade 3 within 4 weeks of start of study medication (CTCAE: Common Terminology Criteria for Adverse Events).
* History or concurrent condition of interstitial lung disease
* Unresolved toxicity higher than CTCAE grade 1 (NCI-CTC version 4.0) attributed to any prior therapy/procedure excluding alopecia. (NCI: National Cancer Institute)
* Prior treatment with PI3K inhibitors
* Systemic corticosteroid therapy (ongoing)
* Hepatitis B or C. All subjects must be screened for hepatitis B and C up to 28 days prior to study drug start using the hepatitis virus panel laboratorial routine. Subjects positive for HBsAg or HBcAb will be eligible if they are negative for HBV-DNA; subjects positive for HCV IgG will be eligible if they are negative for HCV RNA.
* For Part B:

  * Histologically confirmed diagnosis of follicular lymphoma grade 3b or transformed disease and chronic lymphocytic leukemia (CLL)
  * History or concurrent condition of interstitial lung disease or severely impaired pulmonary function
* Excluded medical conditions:

  * Previous or concurrent cancer that is distinct in primary site or histology from indolent B-cell NHL within 5 years prior to treatment start EXCEPT for curatively treated cervical cancer in situ, nonmelanoma skin cancer and superficial bladder tumors [Ta (non-invasive tumor), Tis (carcinoma in situ) and T1 (tumor invades lamina propria)].
  * Hepatitis B or C. All subjects must be screened for hepatitis B and C up to 28 days prior to study drug start using the hepatitis virus panel laboratorial routine. Subjects positive for HBsAg or HBcAb will be eligible if they are negative for HBV-DNA; subjects positive for HCV IgG will be eligible if they are negative for HCV-RNA.
  * Type I or II diabetes mellitus with HbA1c > 8.5% or fasting plasma glucose > 160 mg/dL at screening.
  * Previous or concurrent cancer that is distinct in primary site or histology from indolent B-cell NHL within 5 years prior to treatment start EXCEPT for curatively treated cervical cancer in situ, nonmelanoma skin cancer and superficial bladder tumors [Ta (non-invasive tumor), Tis (carcinoma in situ) and T1 (tumor invades lamina propria)].

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 227 (Actual)
Dates: Start 2012-11-19 (Actual); Primary Completion 2016-06-22 (Actual); Study Completion 2023-05-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (96):
- United States (15):
  - Birmingham, Alabama
  - Gilbert, Arizona
  - Anaheim, California
  - Aurora, Colorado
  - Englewood, Colorado
  - Fort Collins, Colorado
  - Seattle, Florida
  - Louisville, Kentucky
  - Detroit, Michigan
  - Saint Louis Park, Minnesota
  - Westbury, New York
  - Clinton, North Carolina
  - Canton, Ohio
  - San Antonio, Texas
  - Spokane, Washington
- Garran, Australian Capital Territory, Australia
- Linz, Austria
- Belgium (6):
  - Brussels
  - Bruxelles - Brussel
  - Ghent
  - Leuven
  - Turnhout
  - Wilrijk
- Sofia, Bulgaria
- Canada (2):
  - Saint John, New Brunswick
  - Montreal, Quebec
- Finland (4):
  - Helsinki
  - Oulu
  - Tampere
  - Turku
- France (10):
  - Brest
  - Créteil
  - La Roche-sur-Yon
  - Lille
  - Paris
  - Pessac
  - Pierre-Bénite
  - Poitiers
  - Rouen
  - Vandœuvre-lès-Nancy
- Germany (7):
  - München, Bavaria
  - Münster, North Rhine-Westphalia
  - Recklinghausen, North Rhine-Westphalia
  - Mainz, Rhineland-Palatinate
  - Dresden, Saxony
  - Potsdam, State of Berlin
  - Berlin
- Athens, Greece
- Hong Kong (2):
  - Hong Kong
  - Shatin
- Hungary (2):
  - Budapest
  - Kaposvár
- Galway, Ireland
- Israel (3):
  - Petah Tikva
  - Ramat Gan
  - Ẕerifin
- Italy (6):
  - Napoli, Campania
  - Bologna, Emilia-Romagna
  - Rome, Lazio
  - Brescia, Lombardy
  - Milan, Lombardy
  - Turin, Piedmont
- Christchurch, New Zealand
- Poland (2):
  - Gdynia
  - Krakow
- Lisbon, Portugal
- Russia (6):
  - Kemerovo
  - Moscow
  - Nizhny Novgorod
  - Omsk
  - Saint Petersburg
  - Saratov
- Singapore, Singapore
- South Korea (3):
  - Busan, Busan Gwang''yeogsi
  - Seoul, Seoul Teugbyeolsi
  - Seoul
- Spain (6):
  - Majadahonda, Madrid
  - Marbella, Málaga
  - Barcelona
  - Madrid
  - Seville
  - Valencia
- Uddevalla, Sweden
- Turkey (Türkiye) (3):
  - Ankara
  - Istanbul
  - Izmir
- United Kingdom (10):
  - Cambridge, Cambridgeshire
  - Plymouth, Devon
  - Southampton, Hampshire
  - Harrow, London
  - Liverpool, Merseyside
  - Sutton, Surrey
  - Birmingham, West Midlands
  - Leeds
  - Manchester
  - Romford

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.

REFERENCES:
- [Result] Dreyling M, Morschhauser F, Bouabdallah K, Bron D, Cunningham D, Assouline SE, Verhoef G, Linton K, Thieblemont C, Vitolo U, Hiemeyer F, Giurescu M, Garcia-Vargas J, Gorbatchevsky I, Liu L, Koechert K, Pena C, Neves M, Childs BH, Zinzani PL. Phase II study of copanlisib, a PI3K inhibitor, in relapsed or refractory, indolent or aggressive lymphoma. Ann Oncol. 2017 Sep 1;28(9):2169-2178. doi: 10.1093/annonc/mdx289. PMID 28633365
- [Derived] Morcos PN, Moss J, Veasy J, Hiemeyer F, Childs BH, Garmann D. Model-Based Benefit/Risk Analysis for the Copanlisib Intermittent Dosing Regimen. Clin Pharmacol Ther. 2024 May;115(5):1092-1104. doi: 10.1002/cpt.3173. Epub 2024 Jan 16. PMID 38226495
- [Derived] Panayiotidis P, Follows GA, Mollica L, Nagler A, Ozcan M, Santoro A, Stevens D, Trevarthen D, Hiemeyer F, Garcia-Vargas J, Childs BH, Zinzani PL, Dreyling M. Efficacy and safety of copanlisib in patients with relapsed or refractory marginal zone lymphoma. Blood Adv. 2021 Feb 9;5(3):823-828. doi: 10.1182/bloodadvances.2020002910. PMID 33560394
- See also: Click here to find further information and, after study completion, the study results according to Bayer's transparency standards. — https://clinicaltrials.bayer.com/study/16349
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe — http://www.clinicaltrialsregister.eu/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Part A-Study enrolled participants from 41 study centers in 10 countries, between 19 NOV 2012 (first participant first visit [FPFV]) and 13 AUG 2018 (last participant last visit [LPLV]). Part B-Study enrolled participants from 81 study centers in 24 countries, between 04 NOV 2013 (FPFV) and 18 MAY 2023 (LPLV),
Pre-assignment Details: Part A: Overall 125 participants were screened, of them 41 were screened but never assigned to treatment. Total 84 were assigned to treatment. Part B: Overall 213 participants were screened, of them 70 were screened but never assigned to treatment. Total 143 were assigned to treatment, of them 1 was suspected as fraudulent and excluded from analysis sets. Therefore 142 participants were evaluable.
Groups:
- Part A: Indolent NHL/CLL: Participants with indolent Non-Hodgkin's lymphoma/Chronic lymphocytic leukemia [iNHL/CLL] received copanlisib 0.8 milligram per kilogram (mg/kg), maximum 65 mg, intravenous (IV) infusion dosing over 1 hour in 100 milliliter (mL) normal saline solution on Days 1, 8, and 15 of a 28-day treatment cycle until occurrence of progressive disease, as defined in the Report of an International Workshop to Standardize Response Criteria for Non-Hodgkin's Lymphomas by Cheson et al. 1999, clinical progression, unacceptable toxicity, or any other criteria meeting withdrawal from study.
- Part A: Aggressive NHL: Participants with aggressive NHL (aNHL) received copanlisib 0.8 mg/kg, maximum 65 mg, IV infusion dosing over 1 hour in 100 mL normal saline solution on Days 1, 8, and 15 of a 28-day treatment cycle until occurrence of progressive disease, as defined in the Report of an International Workshop to Standardize Response Criteria for Non-Hodgkin's Lymphomas by Cheson et al. 1999, clinical progression, unacceptable toxicity, or any other criteria meeting withdrawal from study.
- Part B: Indolent NHL: Participants with indolent B-cell NHL received copanlisib 60 mg or 0.8 mg/kg, IV infusion dosing over 1 hour in 100 mL normal saline solution on Days 1, 8, and 15 of a 28-day treatment cycle until occurrence of progressive disease, as defined in the Revised Response Criteria for Malignant Lymphoma by Cheson et al., 2007, clinical progression, unacceptable toxicity, or any other criteria meeting withdrawal from study.
Period: Overall Study
Arm/Group | Part A: Indolent NHL/CLL | Part A: Aggressive NHL | Part B: Indolent NHL
Started | 33 | 51 | 142
Completed | 0 | 0 | 0
Not Completed | 33 | 51 | 142
Not completed — Protocol Violation | 0 | 1 | 1
Not completed — AE not associated with clinical disease progression | 13 | 10 | 40
Not completed — AE associated with clinical disease progression | 1 | 3 | 11
Not completed — Sponsor Decision | 0 | 0 | 1
Not completed — Protocol Deviation | 0 | 0 | 1
Not completed — Physician Decision | 1 | 2 | 5
Not completed — Withdrawal by Subject | 1 | 1 | 20
Not completed — Trial closure. | 0 | 0 | 1
Not completed — Switching to other therapy | 0 | 1 | 1
Not completed — Progressive disease - clinical progression | 4 | 10 | 9
Not completed — Progressive disease - radiological progression | 12 | 23 | 50
Not completed — Death | 1 | 0 | 1
Not completed — Other | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS) included all participants assigned to study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part A: Indolent NHL/CLL | Part A: Aggressive NHL | Part B: Indolent NHL | Total
Number analyzed (Participants) | 33 | 51 | 142 | 226
Age, Customized [Number; unit: Participants]
  18 to 90 years | 33 | 51 | 142 | 226
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 22 | 71 | 111
  Male | 15 | 29 | 71 | 115
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 6 | 10
  Not Hispanic or Latino | 21 | 36 | 124 | 181
  Unknown or Not Reported | 10 | 13 | 12 | 35
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 15 | 15
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 25 | 40 | 120 | 185
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 8 | 11 | 7 | 26

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR) Based on Independent Review-Part A
Description: Objective response rate was defined as the proportion of participants with a best response rating of complete response (CR), unconfirmed complete response (CRu) or partial response (PR), based on the Report of an International Workshop to Standardize Response Criteria for non-Hodgkins Lymphomas, Cheson, 1999, as evaluated by the Independent Response Adjudication Committee (IRAC). For chronic lymphocytic leukemia (CLL) patients Hallek criteria (2008) were used and assessed by investigator.
Time Frame: Baseline up to the last patient has completed the 16 weeks of treatment
Population: Per protocol set included all patients treated with study drug and evaluated for ORR and had no major protocol deviation. (In Part A, for CLL patients, there was no independent assessment. Instead, the investigator assessment had been used.)
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Part A: Indolent NHL/CLL | Part A: Aggressive NHL
Number analyzed (Participants) | 32 | 48
percentage of participants | 43.75 [28.73 to 59.68] | 27.08 [16.83 to 39.57]
Statistical Analysis 1: Comparison: Part A: Indolent NHL/CLL; Response rate was statistically compared by exact binomial test if higher than 5%; Test type: Superiority or Other; p = 0.0001, Exact binomial test — 0.0001; Response rate = 45.45, 90% CI 2-sided [30.49 to 61.06]
Statistical Analysis 2: Comparison: Part A: Aggressive NHL; Response rate was statistically compared by exact binomial test if higher than 5%; Test type: Superiority or Other; p = 0.0001, Exact binominal test — 0.0001; P-value was based on the original patients in the aggressive arm (for the first 34 patients), not including the additional recruited patients; Response rate = 27.08, 90% CI 2-sided [16.83 to 39.57]

2. Primary Outcome: ORR Based on Independent Review-Part B
Description: Objective response rate was defined as the proportion of participants with a best response rating of CR or PR, based on the International Working Group Revised response Criteria for Malignant Lymphoma, Cheson 2007.
Time Frame: Baseline up to the last patient has completed the 16 weeks of treatment
Population: FAS included all patients assigned to study treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part B: Indolent NHL
Number analyzed (Participants) | 142
percentage of participants | 59.15 [50.60 to 67.32]
Statistical Analysis 1: Comparison: Part B: Indolent NHL; Response rate was statistically compared by exact binomial test if higher than 40%; Test type: Superiority or Other; p < 0.0001, Exact binominal test — 0.001; Response rate = 59.15, 95% CI 2-sided [50.60 to 67.32]

3. Primary Outcome: ORR Based on Investigator Assessment-Part A
Description: Objective response rate was defined as the proportion of participants with a best response rating of CR, CRu or PR, based on the Report of an International Workshop to Standardize Response Criteria for non-Hodgkins Lymphomas, Cheson, 1999. For CLL patients Hallek criteria (2008) were used and assessed by investigator.
Time Frame: Baseline up to the last patient has completed the 16 weeks of treatment
Population: Per protocol set included all patients treated with study drug and evaluated for ORR and had no major protocol deviation. Patients who were not evaluable for ORR and discontinued due to a drug-related toxicity, death / progression by clinical judgment before disease was re-evaluated and included.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Part A: Indolent NHL/CLL | Part A: Aggressive NHL
Number analyzed (Participants) | 32 | 48
percentage of participants | 46.88 [31.54 to 62.66] | 31.25 [20.35 to 43.97]
Statistical Analysis 1: Comparison: Part A: Indolent NHL/CLL; Response rate was statistically compared by exact binomial test if higher than 5%; Test type: Superiority or Other; p = 0.0001, Exact binominal test — 0.0001; Response rate = 46.88, 90% CI 2-sided [31.54 to 62.66]
Statistical Analysis 2: Comparison: Part A: Aggressive NHL; Response rate was statistically compared by exact binomial test if higher than 5%; Test type: Superiority or Other; p = 0.0001, Exact binominal test — 0.0001; Response rate = 31.25, 90% CI 2-sided [20.35 to 43.97]

4. Primary Outcome: ORR Based on Investigator Assessment-Part B
Description: as for outcome 2
Time Frame: Baseline up to the last patient has completed the 16 weeks of treatment
Population: FAS included all patients assigned to study treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part B: Indolent NHL
Number analyzed (Participants) | 142
percentage of participants | 51.41 [42.88 to 59.87]
Statistical Analysis 1: Comparison: Part B: Indolent NHL; Response rate was statistically compared by exact binomial test if higher than 40%; Test type: Superiority or Other; p = 0.0039, Exact binominal test — 0.01; Response rate = 51.41, 95% CI 2-sided [42.88 to 59.87]

5. Secondary Outcome: Duration of Response (DOR) Based on Independent Review-Part A
Description: DOR was defined as the time from the date of the first observed tumor response of CR or PR (whichever was noted earlier) to first subsequent disease progression (either first progressive disease [PD], first clinical progression or first AE associated with clinical disease progression) or death caused by disease progression, if this death occurred before progression was documented. All deaths were considered as 'caused by disease progression' except deaths with the reason "other" or "AE not related to disease progression. DOR was evaluated only for patients with at least one tumor response of CR, CRu, or PR. Some patients may have had no report of disease progression nor death caused by disease progression until the date of the LPLV. With regards to DOR, these patients were considered as right censored at the date of their last tumor assessment after first observed tumor response.
Time Frame: Baseline up to approximately 6 years
Population: PPS included all patients with study drug administration that were evaluable for objective tumor response and had no major protocol deviation.
  DOR was only evaluated for patients with at least one tumor response of CR, Cru (only for Part A) or PR.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Part A: Indolent NHL/CLL | Part A: Aggressive NHL
Number analyzed (Participants) | 14 | 14
Days | 322 [61 to NA] — NA: Value cannot be estimated due to censored data | NA [61 to NA] — NA: Value cannot be estimated due to censored data

6. Secondary Outcome: DOR Based on Independent Review-Part B
Description: as for outcome 5
Time Frame: Baseline up to approximately 9 years 7 months
Population: FAS included all patients assigned to study treatment. DOR was only evaluated for patients with at least one tumor response of CR, Cru (only for Part A) or PR.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part B: Indolent NHL
Number analyzed (Participants) | 85
Months | 14.9 [9.2 to 22.6]

7. Secondary Outcome: DOR Based on Investigator Assessment-Part A
Description: as for outcome 5
Time Frame: Baseline up to approximately 6 years
Population: as for outcome 5
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Part A: Indolent NHL/CLL | Part A: Aggressive NHL
Number analyzed (Participants) | 15 | 15
Days | 189 [56 to 574] | 190 [112 to NA] — NA: Value cannot be estimated due to censored data

8. Secondary Outcome: DOR Based on Investigator Assessment-Part B
Description: as for outcome 5
Time Frame: Baseline up to approximately 9 years 7 months
Population: as for outcome 6
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part B: Indolent NHL
Number analyzed (Participants) | 78
Months | 11.5 [9.2 to 16.1]

9. Secondary Outcome: Progression Free Survival (PFS) Based on Independent Review-Part A
Description: PFS was defined as the time (in days) from the date of the first treatment to the date of first observed PD (radiological or clinical, or first AE associated with clinical PD, whichever was earlier) or death due to any cause (if death occurred before progression was documented).
Time Frame: Baseline up to approximately 6 years
Population: FAS included all patients assigned to study treatment.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Part A: Indolent NHL/CLL | Part A: Aggressive NHL
Number analyzed (Participants) | 33 | 51
Days | 223 [147 to 546] | 70 [47 to 115]

10. Secondary Outcome: PFS Based on Independent Review-Part B
Description: as for outcome 9
Time Frame: Baseline up to approximately 9 years 7 months
Population: FAS included all patients assigned to study treatment.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part B: Indolent NHL
Number analyzed (Participants) | 142
Months | 11.3 [8.1 to 17.6]

11. Secondary Outcome: PFS Based on Investigator Assessment-Part A
Description: as for outcome 9
Time Frame: Baseline up to approximately 6 years
Population: FAS included all patients assigned to study treatment.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Part A: Indolent NHL/CLL | Part A: Aggressive NHL
Number analyzed (Participants) | 33 | 51
Days | 224 [172 to 419] | 70 [47 to 115]

12. Secondary Outcome: PFS Based on Investigator Assessment-Part B
Description: as for outcome 9
Time Frame: Baseline up to approximately 9 years 7 months
Population: FAS included all patients assigned to study treatment.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part B: Indolent NHL
Number analyzed (Participants) | 142
Months | 10.8 [7.2 to 12.8]

13. Secondary Outcome: Overall Survival (OS)-Part A
Description: OS was defined as the time (in days) from the date of first administration of study treatment to death due to any cause. Patients who were alive at the date of the LPLV were censored at the minimum of the date of LPLV and the last available date of evidence that the patient was still alive.
Time Frame: Baseline up to approximately 6 years
Population: FAS included all patients assigned to study treatment.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Part A: Indolent NHL/CLL | Part A: Aggressive NHL
Number analyzed (Participants) | 33 | 51
Days | 657 [391 to NA] — NA: Value cannot be estimated due to censored data | 211 [140 to 399]

14. Secondary Outcome: OS-Part B
Description: OS was defined as the time (in days) from the date of first administration of study treatment to death due to any cause. OS was defined as the time (in days) from the date of first administration of study treatment to death due to any cause. Patients who were alive at the date of the LPLV were censored at the minimum of the date of LPLV and the last available date of evidence that the patient was still alive.
Time Frame: Baseline up to approximately 9 years 7 months
Population: FAS included all patients assigned to study treatment.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part B: Indolent NHL
Number analyzed (Participants) | 142
Months | 59.1 [36.5 to NA] — NA: Value cannot be estimated due to censored data

15. Secondary Outcome: Functional Assessment of Cancer Therapy - Lymphoma Lymphoma Subscale (FACT-Lym LymS) at Week 16 - Part B
Description: HRQoL assessment was used to describe development of patients with copanlisib by using FACT-Lym questionnaire assessment tool. It contains 42 items (questions) covering HRQoL, common lymphoma symptoms and treatment side-effects. The FACT - General (FACT-G) questionnaire contains 27 items covering 4 core HRQoL subscales: Physical Wellbeing (7 items), Social/Family Wellbeing (7), Emotional Wellbeing (6), and Functional Wellbeing (7). The FACT-Lym also includes an Additional Concerns subscale (15 items) (FACT-Lym LymS), addressing issues typically experienced by lymphoma patients. Some of the issues covered include pain, itching, night sweats, trouble sleeping, fatigue and trouble concentrating. FACT-Lym also asks patients about lumps and swelling, fevers, infections, weight, appetite, emotional stability and treatment. Score range for the FACT-Lym LymS was 0 - 60, higher score represent less symptoms. Here in below table "n" signifies evaluable participants for the respective category.
Time Frame: Baseline up to week 16
Population: FAS included all patients assigned to study treatment. The analysis was performed by using last observation carried forward (LOCF) method.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Part B: Indolent NHL
Number analyzed (Participants) | 141
units on a scale
  Baseline: number analyzed (Participants) | 132
  Baseline | 46.50 [40.50 to 52.00]
  Value at Week 16 | 49.00 [42.00 to 54.00]
Statistical Analysis 1: Comparison: Part B: Indolent NHL; Hodges-Lehmann-estimate was used to calculate change to Week 16 and 95% confidence interval; Test type: Superiority or Other; Hodges-Lehmann-estimate = 1.00, 95% CI 2-sided [0.5 to 2.5]

16. Secondary Outcome: Functional Assessment of Cancer Therapy - Lymphoma (FACT-Lym) Total Score at Week 16 - Part B
Description: HRQoL assessment was used to describe development of patients with copanlisib by using FACT-Lym questionnaire assessment tool. It contains 42 items (questions) covering HRQoL, common lymphoma symptoms and treatment side-effects. The FACT - General (FACT-G) questionnaire contains 27 items covering 4 core HRQoL subscales: Physical Wellbeing (7 items), Social/Family Wellbeing (7), Emotional Wellbeing (6), and Functional Wellbeing (7). The FACT-Lym also includes an Additional Concerns subscale (15 items) (FACT-Lym LymS), addressing issues typically experienced by lymphoma patients. Some of the issues covered include pain, itching, night sweats, trouble sleeping, fatigue and trouble concentrating. FACT-Lym also asks patients about lumps and swelling, fevers, infections, weight, appetite, emotional stability and treatment. FACT-Lym total score range was 0-168, higher score indicates better HRQoL. Here, in the below table "n" signifies evaluable participants for the respective category.
Time Frame: Baseline up to week 16
Population: FAS included all patients assigned to study treatment. The analysis was performed by using last LOCF method.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Part B: Indolent NHL
Number analyzed (Participants) | 141
units on a scale
  Baseline: number analyzed (Participants) | 132
  Baseline | 127.50 [113.75 to 145.75]
  Value at Week 16 | 130.83 [113.33 to 146.50]
Statistical Analysis 1: Comparison: Part B: Indolent NHL; Hodges-Lehmann-estimate was used to calculate change to Week 16 and 95% confidence interval; Test type: Superiority or Other; Hodges-Lehmann-estimate = 0.50, 95% CI 2-sided [-0.7 to 3.2]

ADVERSE EVENTS:
Time Frame: After the first study intervention up to 35 days after the end of study intervention, Part A: approximately 6 years. Part B: approximately 9 years 7 months. Adverse event reporting for the all-cause mortality considers all deaths that occurred at any time during the study before the last contact, Part A: approximately 6 years. Part B: approximately 9 years 7 months.
Arm/Group | Part A: Indolent NHL/CLL | Part A: Aggressive NHL | Part B: Indolent NHL
All-Cause Mortality (participants affected / at risk) | 21/33 | 39/51 | 75/142
Serious Adverse Events (participants affected / at risk) | 16/33 | 31/51 | 81/142
Other Adverse Events (participants affected / at risk) | 33/33 | 50/51 | 138/142
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: Indolent NHL/CLL (N=33) | Part A: Aggressive NHL (N=51) | Part B: Indolent NHL (N=142)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 2 (3) | 3 (3)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 4 (5)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Autoimmune haemolytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Aortic valve incompetence (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 3 (3) | 4 (4)
Gastritis (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Melaena (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 9 (9)
General physical health deterioration (General disorders) | 1 (1) | 4 (4) | 2 (2)
Multiple organ dysfunction syndrome (General disorders) | 0 (0) | 1 (1) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 2 (2)
Gallbladder obstruction (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Bronchopulmonary aspergillosis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Cryptococcosis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 3 (3) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 4 (4) | 4 (5) | 20 (25)
Pneumonia pneumococcal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Progressive multifocal leukoencephalopathy (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 0 (0) | 2 (2) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 2 (2) | 2 (2)
Septic shock (Infections and infestations) | 0 (0) | 1 (1) | 2 (2)
Sinusitis (Infections and infestations) | 1 (1) | 1 (2) | 0 (0)
Tooth abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Rectal abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sinusitis aspergillus (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Coronavirus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Enterocolitis infectious (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Klebsiella bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia fungal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (2)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Pneumocystis jirovecii infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Varicella zoster pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Systemic infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Vascular device infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Afferent loop syndrome (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Biliary-vascular fistula (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1) | 1 (1) | 2 (2)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 7 (9)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Tumour flare (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Porocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0) | 0 (0)
Tumour compression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Disorientation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 1 (1) | 2 (2)
Renal impairment (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 2 (2)
Scrotal swelling (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 6 (8)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dermatitis exfoliative generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Preoperative care (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Circulatory collapse (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Embolism (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Superficial vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: Indolent NHL/CLL (N=33) | Part A: Aggressive NHL (N=51) | Part B: Indolent NHL (N=142)
Anaemia (Blood and lymphatic system disorders) | 11 (21) | 12 (13) | 27 (43)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 8 (16)
Neutropenia (Blood and lymphatic system disorders) | 9 (12) | 15 (25) | 40 (117)
Thrombocytopenia (Blood and lymphatic system disorders) | 3 (3) | 3 (3) | 21 (30)
Vertigo (Ear and labyrinth disorders) | 2 (2) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 4 (6) | 1 (1) | 10 (10)
Abdominal pain upper (Gastrointestinal disorders) | 3 (4) | 3 (3) | 11 (16)
Constipation (Gastrointestinal disorders) | 5 (7) | 8 (11) | 18 (21)
Diarrhoea (Gastrointestinal disorders) | 13 (65) | 21 (39) | 51 (98)
Dry mouth (Gastrointestinal disorders) | 3 (3) | 3 (3) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 (2) | 2 (2) | 5 (5)
Nausea (Gastrointestinal disorders) | 10 (17) | 18 (22) | 33 (45)
Oral pain (Gastrointestinal disorders) | 0 (0) | 3 (3) | 3 (3)
Stomatitis (Gastrointestinal disorders) | 4 (6) | 4 (4) | 14 (24)
Vomiting (Gastrointestinal disorders) | 5 (10) | 5 (7) | 20 (25)
Asthenia (General disorders) | 8 (13) | 6 (6) | 11 (14)
Chest pain (General disorders) | 1 (1) | 3 (4) | 2 (2)
Chills (General disorders) | 2 (2) | 1 (1) | 12 (13)
Fatigue (General disorders) | 16 (20) | 14 (15) | 36 (41)
Influenza like illness (General disorders) | 2 (2) | 2 (2) | 6 (6)
Mucosal inflammation (General disorders) | 4 (5) | 6 (8) | 10 (17)
Oedema peripheral (General disorders) | 3 (7) | 2 (2) | 12 (14)
Pyrexia (General disorders) | 10 (14) | 8 (22) | 35 (54)
Bronchitis (Infections and infestations) | 4 (10) | 5 (8) | 16 (22)
Conjunctivitis (Infections and infestations) | 4 (4) | 1 (2) | 6 (9)
Cystitis (Infections and infestations) | 4 (5) | 1 (1) | 1 (1)
Herpes zoster (Infections and infestations) | 2 (2) | 1 (1) | 3 (4)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 3 (6) | 4 (5)
Nasopharyngitis (Infections and infestations) | 1 (2) | 2 (2) | 9 (16)
Oral candidiasis (Infections and infestations) | 0 (0) | 3 (3) | 6 (7)
Pneumonia (Infections and infestations) | 3 (3) | 2 (2) | 12 (14)
Rhinitis (Infections and infestations) | 1 (1) | 1 (1) | 9 (13)
Sinusitis (Infections and infestations) | 1 (1) | 2 (4) | 10 (13)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 2 (2) | 22 (45)
Urinary tract infection (Infections and infestations) | 6 (6) | 7 (7) | 7 (10)
Oral herpes (Infections and infestations) | 1 (2) | 2 (2) | 9 (13)
Procedural pain (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 2 (2)
Blood creatinine increased (Investigations) | 1 (1) | 4 (5) | 6 (6)
Blood glucose increased (Investigations) | 2 (5) | 0 (0) | 2 (42)
Eosinophil count increased (Investigations) | 2 (2) | 1 (1) | 0 (0)
Lipase increased (Investigations) | 2 (4) | 2 (2) | 8 (9)
Neutrophil count decreased (Investigations) | 3 (15) | 1 (2) | 7 (19)
Platelet count decreased (Investigations) | 5 (5) | 4 (4) | 13 (16)
Weight decreased (Investigations) | 0 (0) | 2 (2) | 9 (9)
White blood cell count decreased (Investigations) | 1 (1) | 0 (0) | 8 (8)
Hyperglycaemia (Metabolism and nutrition disorders) | 21 (88) | 27 (55) | 71 (515)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (3) | 5 (5) | 11 (11)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (3) | 10 (11)
Hypophosphataemia (Metabolism and nutrition disorders) | 2 (2) | 4 (4) | 4 (10)
Decreased appetite (Metabolism and nutrition disorders) | 5 (6) | 7 (8) | 15 (15)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (6) | 5 (5) | 14 (15)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (4) | 4 (4) | 14 (22)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 7 (10) | 3 (5) | 12 (17)
Dizziness (Nervous system disorders) | 3 (4) | 3 (4) | 4 (5)
Headache (Nervous system disorders) | 7 (9) | 9 (12) | 14 (22)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 3 (3) | 6 (6)
Paraesthesia (Nervous system disorders) | 3 (3) | 1 (1) | 4 (5)
Somnolence (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Taste disorder (Nervous system disorders) | 2 (2) | 1 (1) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 3 (3) | 4 (5)
Insomnia (Psychiatric disorders) | 0 (0) | 3 (3) | 8 (8)
Dysuria (Renal and urinary disorders) | 2 (2) | 0 (0) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (13) | 6 (6) | 27 (45)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 4 (4) | 11 (11)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 4 (4)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (4) | 3 (3) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0) | 4 (5)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3) | 10 (12)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (3) | 4 (5)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 15 (20)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3) | 7 (10)
Eczema (Skin and subcutaneous tissue disorders) | 3 (4) | 2 (2) | 4 (10)
Erythema (Skin and subcutaneous tissue disorders) | 3 (3) | 3 (3) | 2 (3)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3) | 3 (5) | 14 (37)
Rash (Skin and subcutaneous tissue disorders) | 5 (6) | 6 (8) | 14 (31)
Hypertension (Vascular disorders) | 23 (94) | 24 (82) | 42 (330)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Contract Partners (PI) shall provide to Bayer any proposed publication or oral presentation relating to the Study or the Results ("Publication") at least sixty (60) days prior to the intended submission or presentation of the Publication in order to allow Bayer to review it. If Bayer does not notify PI within forty-five (45) days of Bayer's receipt of the intended Publication, PI shall remind Bayer. If Bayer does not provide any comments within the sixty day period, PI shall be free to publish.